CLINICAL TRIAL: NCT00350714
Title: Validation of a Breath Test for Assessment of Liver Fibrosis in Patients With Chronic Hepatitis C Viral Infection
Brief Title: BreathID Multi-center HCV Liver Breath Test Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to FDA comments, protocol changed; new trial will be proposed shortly
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Baylor College of Medicine (Other); Virginia Commonwealth University (Other); Hadassah Medical Organization (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Dr. Scott Friedman, Mouont Sinai School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MBVH-0706
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis C
Keywords: HCV (Hepatitis C Virus); MBT (Methacetin Breath Test); Hepatitis C Virus Patients
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBT (Experimental): C13 methacetin dissolved in water to be ingested after breath baseline collected. Metabolism to measured in real time.
  Interventions: Other: MBT and BreathID

INTERVENTIONS:
Other: MBT and BreathID — 75 mg methacetin (c13 labelled) dissolved in 150 cc water ingested and breath collected before and after ingestion.

SUMMARY:
The goal of this study is to validate the BreathID 13C-methacetin breath test (MBT) as a non-invasive simple-to-use metabolic test, which could be utilized to detect severe liver fibrosis (>2 in METAVIR) in patients with chronic HCV liver disease.The test is a breath-test using a free-standing device (BreathID®) that measures metabolization of a 13C-labeled substrate (13C-methacetin) in real time.

DETAILED DESCRIPTION:
Percutaneous liver biopsy has been utilized for decades to assess the severity of chronic HCV liver disease. During this procedure a core sample of liver is obtained and examined histologically for the presence of inflammation, fibrosis and other features characteristic of specific liver disorders. Several grading systems have been developed over the past 2 decades to quantify the overall severity of the liver biopsy specimen. Although liver biopsy is the gold standard by which to assess liver disease severity, the procedure has significant limitations. Liver biopsy is a costly, invasive procedure with risks for morbidity and mortality and may cause some discomfort to the patient. Percutaneous liver biopsy is associated with potential complications, including bleeding (1%-3%), pain (20%-30%), bile peritonitis (<1%), pneumothorax (<1%), punctured viscera (<1%), and death. In addition, liver biopsy and examination of liver histology is subject to sampling variation and the manner by which these findings are evaluated and reported by individual pathologists.

Breath testing with 13C-labeled substrates provide a safe, non-invasive means for evaluating hepatic metabolism that is correlated with liver histology. 13C is a stable, non-radioactive isotope, which can by incorporated into a specific location within a test substrate so that it would be released when the compound is metabolized by the liver. Ideally, the 13C-compound would need to be administered orally, rapidly absorbed, exclusively metabolized by the liver metabolism and 13C would be measured in exhaled breath within 20-30 minutes. Hepatic metabolism of the compound is assessed by measuring the ratio of 13C/12C in exhaled breath. The ability to detect, differentiate and quantify 13C and 12C in exhaled CO2 has been greatly facilitated by the recent development of the BreathID® collection system and analyzer unit.

The compound selected for this study will be 13C-methacetin. Methacetin meets all of the qualifications for an excellent substrate for liver breath tests. It is a non-toxic small molecule. 13C can be synthesized into a key location within this agent. It can be administered orally in solution. It is rapidly absorbed and metabolized by hepatic microsomes and this process releases CO2 as a by-product in exhaled breath. No reports of any complications or side effects using this substance have been reported.

13C-methacetin is rapidly absorbed and metabolized by healthy liver cells into acetaminophen and 13CO2. The resultant CO2 can be measured in the exhaled breath. The amount of metabolized methacetin indicates the capability of the liver to accomplish one of its main physiological tasks and has been shown to correlate with liver fibrosis and cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

i. Patients with a confirmed diagnosis of Chronic HCV only : ii. Patients for whom a liver biopsy has been performed within the last 90 days or who will undergo a liver biopsy within the time frame of the study.

Exclusion Criteria:

i. Severe congestive heart failure. ii. Severe pulmonary hypertension. iii.Chronic renal insufficiency defined by a serum creatinine above the limits of normal. iv. Uncontrolled diabetes mellitus (need definition).v.Any autoimmune disorder, which is currently being treated with prednisone or any other immune suppressive medication. vi.Proven or suspected hepatocellular carcinoma. vii. Previous surgical bypass surgery for morbid obesity viii.Extensive small bowel resection. ix.Patients currently receiving total parenteral nutrition x.Recipients of any organ transplant. xi.Other co-existent liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Correlation of Breath Test (MBT) to Fibrosis | 12 months
  13 C Lebeled substrate is metabolized by Liver and reflects liver function. It is hypothesized that this correlated to liver fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Doug Dieterich, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; John M Vierling, MD, Principal Investigator — Baylor College of Medicine; Mitchell Shiffman, MD, Principal Investigator — Virginia Commonwealth University; Maya Margalit, MD, Principal Investigator — Hadassah Medical Organization; Douglas M. Heuman, M.D., Principal Investigator — U.S. Dept. of Veteran Affairs, Hunter Holmes McGuire Medical Center
Locations (5):
- United States (4):
  - Mount Sinai School of Medicine, New York, New York
  - Baylor College of Medicine, Houston, Texas
  - U.S. Dept. of Veteran Affairs, Hunter Holmes McGuire Medical Center, Richmond, Virginia
  - Virginia Commonwealth Univeristy, Richmond, Virginia
- Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Result] O. Goetze; N. Selzner; A. Grau; M. Fried; T. Gerlach; B. Muellhaupt 13C-Methacetin Breath Test by Online Molecular Correlation Spectroscopy Compared to APRI and Liver Biopsy for the Assessment of Fibrosis in Chronic Hepatitis C , S1047. Abstarct presented at DDW 2006
- See also: Website of BreathID whose device will be used in this study — http://www.breathid.com